CLINICAL TRIAL: NCT04448522
Title: A Multicenter Randomized Controlled Trial Comparing Reduced Dose With Regular Dose Intensity-modulated Radiotherapy for Chemotherapy Sensitive Stage II-III Nasopharyngeal Carcinoma
Brief Title: Reduced vs Conventional Dosage Intensity-modulated Radiotherapy for Chemotherapy-sensitive Stage II-III Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: National Cancer Centre, Singapore (Other); Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); Zhongshan People's Hospital, Guangdong, China (Other); Yuebei People's Hospital (Other); Wuzhou Red Cross Hospital (Other)
Responsible Party: Principal Investigator, Ming-Yuan Chen, Proffessor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-MYC-2020-1201
Record Dates: First submitted 2020-06-24; First posted 2020-06-26 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Nasopharyngeal Carcinoma; Radiotherapy; Chemotherapy
Keywords: Nasopharyngeal carcinoma; intensity-modulated radiotherapy; chemotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduced dosage IMRT group (Experimental): 3 cycles of gemcitabin and cisplatin induction chemotherapy plus concurrent cheomtherapy with IMRT dosage of 63.6 Gy
  Interventions: Radiation: reduced dosage IMRT
- Conventional dosage IMRT group (Active Comparator): 3 cycles of gemcitabin and cisplatin induction chemotherapy plus concurrent cheomtherapy with IMRT dosage of 69.96 Gy
  Interventions: Radiation: conventional dosage IMRT

INTERVENTIONS:
Radiation: reduced dosage IMRT — 1. Gemcitabine plus cisplatin induction chemotherapy: gemcitabine is injected intravenously at the dose of 1000 mg/m2 on the 1st and 8th day (within 30 minutes) for 3 cycles; cisplatin is injected intravenously at the dose of 80 mg/m2 on the 1st day, for 3 cycles. 1 cycles per 3 weeks.
  2. Concurrent cisplatin chemotherapy: cisplatin is given at a dose of 100 mg/m2 via a continuous intravenous infusion during radiotherapy and starts on the 1st day of radiotherapy for 2 cycles. 1 cycles per 3 weeks.
  3. IMRT: PTVnx：63.6Gy/30Fr/2.12Gy; PTVnd：63.6Gy/30Fr/2.12Gy; PTV1：54Gy/30Fr/1.8Gy; PTV2：49.2Gy/30Fr/1.64Gy
  Arms: Reduced dosage IMRT group
Radiation: conventional dosage IMRT — 1. Gemcitabine plus cisplatin induction chemotherapy: gemcitabine is injected intravenously at the dose of 1000 mg/m2 on the 1st and 8th day (within 30 minutes) for 3 cycles; cisplatin is injected intravenously at the dose of 80 mg/m2 on the 1st day, for 3 cycles. 1 cycles per 3 weeks.
  2. Concurrent cisplatin chemotherapy: cisplatin is given at a dose of 100 mg/m2 via a continuous intravenous infusion during radiotherapy and starts on the 1st day of radiotherapy for 2 cycles. 1 cycles per 3 weeks.
  3. IMRT: PTVnx：69.96Gy/33Fr/2.12Gy; PTVnd：69.96Gy/33Fr/2.12Gy; PTV1：59.4Gy/33Fr/1.8Gy; PTV2：54Gy/33Fr/1.64Gy
  Arms: Conventional dosage IMRT group

SUMMARY:
Through multicenter, open-label, randomised clinical trials, we intend to demonstrate that radiotherapy with reduced dose could significantly reduce the incidence of radiotherapy toxicities, improve the quality of life of patients while ensuring the tumor control rates for NPC patients staged as II-III who are sensitive to induction chemotherapy (imaging evaluation of CR/PR and EBV DNA copy number decreased to 0 copies/mL after induction chemotherapy)

DETAILED DESCRIPTION:
Through multicenter, open-label, randomised clinical trials, patients with NPC staged as II-III with CR/PR according to RECIST criteria and EBV DNA decreased to 0 copies/mL after 3 cycles of GP induction chemotherapy will be randomized into experimental group to receive IMRT of reduced dose (prescribed dose, 63.6 Gy, 2.12 Gy per fractions, 30 fractions) and control group to receive IMRT of conventional dose (prescribed dose, 69.96 Gy, 2.13 Gy per time, 33 fractions). Two cycles of cisplatin chemotherapy will be performed during IMRT. The efficacy, toxicity, and quality of life of patients between the two groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed non-keratinizing nasopharyngeal carcinoma (differentiated or undifferentiated type, i.e., WHO type II or type III).
2. Staged as T1-3N1-2M0, T2-3N0M0 (stage II-III) at diagnosis (according to the 8th AJCC edition).
3. Aged between 18-70 years.
4. Karnofsky scale (KPS)≥70.
5. Normal bone marrow function.
6. Evaluated as PR or CR after 3 cycles of GP induction chemotherapy.
7. EBV DNA copy number decreased to 0 copies/mL after 3 cycles of GP induction chemotherapy.
8. Normal liver and kidney function:

   1. total bilirubin, AST and ALT levels of no more than 2.5 times the upper normal limit;
   2. creatinine clearance rate of at least 60 mL/min or creatinine of no more than 1.5 times the upper normal limit.
9. Given written informed consent.

Exclusion Criteria:

1. Histologically confirmed keratinized squamous cell carcinoma (WHO type I) or basal squamous cell carcinoma.
2. Recurrent or metastatic nasopharyngeal carcinoma.
3. Evaluated as SD or PD after 3 cycles of GP induction chemotherapy.
4. EBV DNA copy number of more than 0 copies/mL after 3 cycles of GP induction chemotherapy.
5. Pregnancy or lactation (Pregnancy tests should be considered for women in childbearing age, and effective contraception should be emphasized during treatment.)
6. Other invasive malignant diseases in the past, other than cured basal cell skin carcinoma, squamous cell carcinoma, cervical carcinoma in situ.
7. Primary and regional lesions have been treated with chemotherapy or surgery (except diagnostic purpose)
8. Any severe disease, which may cause unacceptable risk factors or affect compliance with the trial, for example, unstable heart disease requiring treatment, kidney disease, chronic hepatitis, poorly controlled diabetes (fasting blood glucose > 1.5×ULN), and mental illness.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Estimated)
Dates: Start 2020-08-18 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival (PFS) | 3 years
  Defined as time from randomization to locoregional or distant metastasis relapse or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall Survival (OS) | 3 years
  Defined as the time interval from randomization to death due to any cause.
Distant Metastasis-Free Survival (DMFS) | 3 years
  Defined as the time interval from randomisation to the date of first distant metastases.
Locoregional Relapse-Free Survival (LRRFS) | 3 years
  Defined as the time from randomisation to the date of first locoregional relapse.
Incidence of treatment related acute complications | up to 1 years
  The proportion of patients with treatment related acute complications according to NCI-CTC5.0 criteria and RTOG criteria.
Incidence of treatment related late complications | up to 3 years
  The proportion of patients with treatment related late complications according to NCI-CTC5.0 criteria and RTOG criteria.
Score of survival quality according to the EORTC Quality of Life Questionnaire (QLQ)-C30 (V3.0) | up to 3 years
  Score of survival quality according to the EORTC Quality of Life Questionnaire (QLQ)-C30 (V3.0) before treatment, during treatment, after treatment.
Score of survival quality according to the EORTC Quality of Life Questionnaire Head and Neck (The QLQ-H&N35) | up to 3 years
  Score of survival quality according to the EORTC Quality of Life Questionnaire Head and Neck (The QLQ-H&N35) before treatment, during treatment, after treatment.

CONTACTS AND LOCATIONS:
Locations (6):
- China (5):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Cancer Center of Guangzhou Medical University, Guangzhou, Guangdong
  - Yuebei People's Hospital, Shaoguan, Guangdong
  - Zhongshan People's Hospital, Zhongshan, Guangdong
  - Wuzhou Red Cross Hospital, Wuzhou, Guangxi
- National Cancer Centre Singapore, Singapore, Singapore